CLINICAL TRIAL: NCT06638086
Title: Effectiveness Of Intravenous Vs Rectal Acetaminophen For Pain Management In Post Operative Neonates; A Randomised Controlled Trial
Brief Title: Effectiveness Of Intravenous Vs Rectal Acetaminophen For Pain Management In Post Operative Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Hasnain Aslam, Principal Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMU-RRF-SUR-008-23
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pain Score Reduction; Effectiveness of Acetaminophen; Postoperative Pain Management in Neonates; Rescue Analgesia; Neonatal Patient
Keywords: Neonatal analgesia protocols; Neonatal care; Pain score reduction; Neonatal pain management; Acetaminophen in neonates; Pediatric surgery pain relief
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: The interventional study model for this article is a Parallel Assignment model.
  In this study, neonates are randomly assigned to one of two groups: one group receives intravenous (IV) acetaminophen, and the other group receives rectal acetaminophen. The outcomes, such as the need for rescue analgesia, time to rescue analgesia, and reduction in pain scores, are then compared between these two parallel groups to assess the effectiveness of the different administration routes for managing postoperative pain in neonates.
Masking Description: The primary investigator collects and analyzes the data using self-designed questionnaires. Typically, in such studies, the intervention (route of acetaminophen) would be known to the healthcare providers administering. Therefore, masking of the participants and providers might not be feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Per-rectal group (Experimental): These neonates received Acetaminophen per rectally at dose of 40 mg/kg.
  Interventions: Drug: Acetaminophen Suppositories
- Intra-vanous group (Active Comparator): These neonates received intravenous Acetaminophen at dose of 15 mg/kg.
  Interventions: Drug: Acetaminophen Injection

INTERVENTIONS:
Drug: Acetaminophen Suppositories — Per rectal suppositories
  Other Names: Napa Suppositories
  Arms: Per-rectal group
Drug: Acetaminophen Injection — Intra-venous injection
  Other Names: Provase
  Arms: Intra-vanous group

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of intravenous (IV) versus rectal acetaminophen for postoperative pain management in neonates. The study includes postoperative term neonates who require analgesia for at least 12 hours. The main questions the study seeks to answer are:

Does IV acetaminophen provide better pain relief compared to rectal administration in neonates? What is the time to rescue analgesia and the efficacy of pain score reduction between these two routes? The study compares 32 neonates receiving IV acetaminophen to 32 neonates administered rectal acetaminophen. Both routes are administered at equivalent bioavailable doses to ensure a fair comparison.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the comparative effectiveness of intravenous (IV) versus rectal administration of acetaminophen for managing postoperative pain in neonates. Neonates, due to their limited physiological reserves and underdeveloped metabolic systems, require precise pain management strategies to prevent potential developmental delays or adverse effects. Acetaminophen, a commonly used analgesic in neonatal care, is metabolized primarily by the liver and excreted via the kidneys. However, its pharmacokinetics vary significantly based on the route of administration, making it important to evaluate which method offers more reliable pain relief.

The study includes 64 term neonates who underwent surgery and are expected to require pain relief for at least 12 hours. Preterm and preoperative neonates are excluded. The neonates were randomized into two groups: one receiving acetaminophen intravenously (15 mg/kg) and the other rectally (40 mg/kg), ensuring similar concentrations at the effect site.

Key variables include rescue analgesia requirements, time to rescue analgesia, and changes in pain scores. Pain relief efficacy is measured by pain score changes, and any need for additional analgesia is recorded.

This study will provide valuable insights into the optimal route for administering acetaminophen in neonates.

ELIGIBILITY:
Inclusion Criteria:

* All post-operative neonates requiring acetaminiphen as analgesia.

Exclusion Criteria:

* All neonates requiring any other kind of Pain relief medication (Nerve block or local analgesia)
* All neonates in neonatal ICU
* All neonates with central venous line in place
* All neonates that are on ventilatory support

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
change in pain score | 0 to 6 hours
  "Bernese Pain Scale for Neonates" will be used consisting of total score of 27
Time for rescue analgesia | 0 to 6 hours
  time will be measured and compared

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza Chaudhry, MBBS, MS, Study Director — Rawalpindi Medical College; Mudassar Fiaz Gondal, MBBS, MS, Study Chair — Rawalpindi Medical College; Hasnain Aslam, MBBS, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Department of Pediatric Surgery,Holy Family Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grunau RE, Whitfield MF, Petrie-Thomas J, Synnes AR, Cepeda IL, Keidar A, Rogers M, Mackay M, Hubber-Richard P, Johannesen D. Neonatal pain, parenting stress and interaction, in relation to cognitive and motor development at 8 and 18 months in preterm infants. Pain. 2009 May;143(1-2):138-46. doi: 10.1016/j.pain.2009.02.014. PMID 19307058
- [Result] Cuzzolin L, Antonucci R, Fanos V. Paracetamol (acetaminophen) efficacy and safety in the newborn. Curr Drug Metab. 2013 Feb;14(2):178-85. PMID 22935063
- [Result] Duggan ST, Scott LJ. Intravenous paracetamol (acetaminophen). Drugs. 2009;69(1):101-13. doi: 10.2165/00003495-200969010-00007. PMID 19192939
- [Result] Walls L, Baker CF, Sarkar S. Acetaminophen-induced hepatic failure with encephalopathy in a newborn. J Perinatol. 2007 Feb;27(2):133-5. doi: 10.1038/sj.jp.7211641. PMID 17262050
- [Result] Hansen TG, O'Brien K, Morton NS, Rasmussen SN. Plasma paracetamol concentrations and pharmacokinetics following rectal administration in neonates and young infants. Acta Anaesthesiol Scand. 1999 Sep;43(8):855-9. doi: 10.1034/j.1399-6576.1999.430813.x. PMID 10492416
- [Result] Anderson BJ, van Lingen RA, Hansen TG, Lin YC, Holford NH. Acetaminophen developmental pharmacokinetics in premature neonates and infants: a pooled population analysis. Anesthesiology. 2002 Jun;96(6):1336-45. doi: 10.1097/00000542-200206000-00012. PMID 12170045
- [Result] Capici F, Ingelmo PM, Davidson A, Sacchi CA, Milan B, Sperti LR, Lorini L, Fumagalli R. Randomized controlled trial of duration of analgesia following intravenous or rectal acetaminophen after adenotonsillectomy in children. Br J Anaesth. 2008 Feb;100(2):251-5. doi: 10.1093/bja/aem377. PMID 18211998